CLINICAL TRIAL: NCT03201523
Title: Evaluation of a Socio-ecological Cardiovascular Disease Prevention Intervention for Ultra-Orthodox Jewish Hasidic Women Using a Participatory Approach
Brief Title: Evaluation of a Socio-ecological Cardiovascular Disease Prevention Intervention for Ultra-Orthodox Jewish Hasidic Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Donna R Zwas, Director of Linda Joy Pollin Cardiovascular Wellness Center for Women, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 465BLZ-HMO-CTIL
Record Dates: First submitted 2017-03-06; First posted 2017-06-28 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Cardiovascular Diseases; Health Behavior
Keywords: Community-based Intervention; Socio-ecological Model; Participatory Approach; Ultra-Orthodox Jewish women
MeSH Terms: conditions — Cardiovascular Diseases; Health Behavior

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental, pre-post study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Community members will be exposed to multiple interventions designed through the participatory approach, integrating the socio-ecological model.
  Interventions: Other: Socio-ecologial, community-based intervention

INTERVENTIONS:
Other: Socio-ecologial, community-based intervention — Intervention components will include a health newsletter, health workshops, community evening/health project registration, lay leader training, neighborhood exercise groups, community walking programs with pedometers, healthy cooking contest, and school health promotion activities.

SUMMARY:
The purpose of this research study is to design, implement, and evaluate a community level, socio-ecological based CVD prevention intervention using a participatory approach for women in a homogeneous ultra-Orthodox Jewish Hasidic community in Israel. A quasi-experimental, pre-post study design will be utilized, where all community participants will be exposed to intervention components. Pre and post samples will be selected through randomized cluster sampling of pre-existing community groups. It is hypothesized that ultra-Orthodox Jewish Hasidic women exposed to this community intervention will have improved healthy eating behaviors, reduced unhealthy eating behaviors, increased engagement in physical activity and sleep, and reduced risk for obesity (weight, BMI).

DETAILED DESCRIPTION:
The purpose of this research study is to design, implement, and evaluate a community level, socio-ecological based CVD prevention intervention using a participatory approach for women in a homogeneous ultra-Orthodox Jewish Hasidic community in Israel. A quasi-experimental, pre-post study design will be utilized, where all community participants will be exposed to intervention components. Pre and post samples will be selected through randomized cluster sampling of pre-existing community groups (n=239 ). Intervention components will be designed through qualitative and quantitative data collection (focus groups, interviews, and questionnaires) from the target population and implementation will be conducted in partnership with community organizations. Intervention components will include a health newsletter, health workshops, community evening/health project registration, lay leader training, neighborhood exercise groups, community walking programs with pedometers, healthy cooking contest, and school health promotion activities. It is hypothesized that ultra-Orthodox Jewish Hasidic women exposed to this community intervention will have improved healthy eating behaviors, reduced unhealthy eating behaviors, increased engagement in physical activity and sleep, and reduced risk for obesity (weight, BMI).

ELIGIBILITY:
Inclusion Criteria:

* Hebrew, English, or Yiddish speaker
* Ultra-Orthodox Jewish Hasidic woman in the targeted community

Exclusion Criteria:

* None

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 239 (Estimated)
Dates: Start 2013-11-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Eating behaviors | One year following project completion (4 years later)
  Eating behaviors will be assesses through self report of specific food item consumption via questionnaire
Engagement in physical activity | One year following project completion (4 years later)
  Engagement in physical activity will be assesses through self report of minutes engaged in vigorous and moderate physical activity via questionnaire as well as pedometer step count where relevant
Reduced risk for obesity (weight, BMI). | One year following project completion (4 years later)
  Self report of BMI
Hours of sleep | One year following project completion (4 years later)
  Hours of sleep will be assesses through self report of average hours slept via questionnaire

SECONDARY OUTCOMES:
General Health Self Efficacy | One year following project completion (4 years later)
  General Health Self Efficacy will be assessed via Ralph Schwarzer's General Health Self Efficacy self report scale, culturally adapted to the population
Spiritual Health Locus of Control | One year following project completion (4 years later)
  Spiritual Health Locus of Control will be measured through Holt's Spiritual Health Locus of Control scale, culturally adapted to the population
self perceived health status | One year following project completion (4 years later)
  self perceived health status will be assessed through self report questionnaire
Cardiovascular disease knowledge | One year following project completion (4 years later)
  Cardiovascular disease knowledge will be assesses through self report questionnaire based on the American Heart Association's knowledge survey items
Stages of Change for targeted health behaviors | One year following project completion (4 years later)
  Stages of Change for targeted health behaviors will be assesses through self report questionnaire
health parameters of local population | 3 years prior to intervention, 2 years after intervention.
  data will be retrieved from local health plans including lipid profile, weight and hemoglobin a1c

CONTACTS AND LOCATIONS:
Overall Officials: Donna Zwas, MD, MPH, Principal Investigator — Hadassah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oguma Y, Shinoda-Tagawa T. Physical activity decreases cardiovascular disease risk in women: review and meta-analysis. Am J Prev Med. 2004 Jun;26(5):407-18. doi: 10.1016/j.amepre.2004.02.007. PMID 15165657
- [Background] Barton P, Andronis L, Briggs A, McPherson K, Capewell S. Effectiveness and cost effectiveness of cardiovascular disease prevention in whole populations: modelling study. BMJ. 2011 Jul 28;343:d4044. doi: 10.1136/bmj.d4044. PMID 21798967
- [Background] McLeroy KR, Bibeau D, Steckler A, Glanz K. An ecological perspective on health promotion programs. Health Educ Q. 1988 Winter;15(4):351-77. doi: 10.1177/109019818801500401. PMID 3068205
- [Background] Macaulay AC, Commanda LE, Freeman WL, Gibson N, McCabe ML, Robbins CM, Twohig PL. Participatory research maximises community and lay involvement. North American Primary Care Research Group. BMJ. 1999 Sep 18;319(7212):774-8. doi: 10.1136/bmj.319.7212.774. No abstract available. PMID 10488012
- [Background] Horowitz CR, Robinson M, Seifer S. Community-based participatory research from the margin to the mainstream: are researchers prepared? Circulation. 2009 May 19;119(19):2633-42. doi: 10.1161/CIRCULATIONAHA.107.729863. PMID 19451365
- [Background] Hu FB, Willett WC. Optimal diets for prevention of coronary heart disease. JAMA. 2002 Nov 27;288(20):2569-78. doi: 10.1001/jama.288.20.2569. PMID 12444864